CLINICAL TRIAL: NCT00866606
Title: An Evaluation Of The Safety And Efficacy Of On-Demand Treatment With BeneFIX (Nonacog Alfa, Recombinant Factor IX) In Chinese Subjects With Hemophilia B
Brief Title: Study Evaluating On-Demand Treatment With BeneFIX In Chinese Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3090A1-3305; B1821004
Record Dates: First submitted 2009-03-19; First posted 2009-03-20 (Estimated); Results first posted 2011-01-04 (Estimated); Last update posted 2011-04-05 (Estimated); Status verified 2011-04

CONDITIONS: Hemophilia B
Keywords: On-demand treatment; Hemostatic efficacy; Factor IX activity; Factor IX recovery; Factor IX inhibitor; Chinese
MeSH Terms: conditions — Hemophilia B | interventions — Factor IX

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Benefix (Experimental): Subjects received on-demand treatments with BeneFIX over a 6-month (calendar day) period.
  Interventions: Biological: Benefix

INTERVENTIONS:
Biological: Benefix — BeneFIX for on-demand treatment of bleeding episodes were according to investigator prescription. FIX recovery was assessed by determining the FIX activity (FIX:C) levels in individual subjects. BeneFIX dosage for recovery assessments: single 75 IU/kg (±5 IU/kg) IV bolus infusion.

SUMMARY:
This study will evaluate the safety and efficacy of on-demand treatment with BeneFIX in Chinese hemophilia B subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subjects equal or more than 6 years of age with mild, moderate or severe hemophilia B (FIX activity: more than 5%, 1-5%, or less than 1%, respectively)
* Subjects with previous exposure to FIX replacement therapy
* If HIV positive, documented CD4 count more than 200/µL within 6 months of study entry

Exclusion Criteria:

* Diagnosed with any bleeding disorder in addition to hemophilia B
* Current FIX inhibitor or history of FIX inhibitor (defined as >ULN of the reporting laboratory)
* Subject has no history of exposure to FIX products (previously untreated patient [PUP])
* Subject is currently utilizing primary FIX prophylaxis
* Subjects anticipating elective surgery that may be planned to occur in the 6 months following study entry
* Treated with immunomodulatory therapy within 30 days prior to study entry or planned use for the duration of their study participation
* Participated in another investigational drug or device study within 30 days prior to study entry or planned participation for the duration of their study participation
* Subjects with a known hypersensitivity to hamster protein
* Significant hepatic or renal impairment (ALT and AST >5 x ULN, bilirubin >2 mg/dL or serum creatinine >1.25 x ULN)
* Prothrombin Time >1.5 x ULN
* Platelet count <80,000/µL
* Pregnant or breastfeeding women
* Unwilling or unable to follow the terms of the protocol
* Any condition which may compromise the subject's ability to comply with and/or perform study-related activities or that poses a clinical contraindication to study participation, in the opinion of the Investigator or Sponsor

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2009-02; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (6):
- China (6):
  - Pfizer Investigational Site, Guangzhou, Guangzhou
  - Pfizer Investigational Site, Suzhou, Jiangsu
  - Pfizer Investigational Site, Tianjin, Tianjin Municipality
  - Pfizer Investigational Site, Hangzhou, Zhejiang
  - Pfizer Investigational Site, Beijing
  - Pfizer Investigational Site, Shanghai

REFERENCES:
- [Derived] Yang R, Zhao Y, Wang X, Sun J, Jin J, Wu D, Charnigo R, O'Brien A, Zhong Z, Rendo P. Evaluation of the safety and efficacy of recombinant factor IX (nonacog alfa) in minimally treated and previously treated Chinese patients with haemophilia B. Haemophilia. 2012 Sep;18(5):e374-8. doi: 10.1111/j.1365-2516.2012.02907.x. Epub 2012 Jul 9. No abstract available. PMID 22776196
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3090A1-3305&StudyName=Study%20Evaluating%20On-Demand%20Treatment%20With%20BeneFIX%20In%20Chinese%20Subjects

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled in six centers in China.
Groups:
- BeneFactor IX (BeneFIX): Participants received on-demand treatments with BeneFIX according to investigator's prescription over a 6-month (calendar day) period. A single 75 International Unit (IU)/kg (±5 IU/kg) intravenous (IV) bolus infusion of BeneFIX was given for recovery assessments. All BeneFIX administrations occurred in the clinic (hospital).
Period: Overall Study
Arm/Group | BeneFactor IX (BeneFIX)
Started | 35
Completed | 31
Not Completed | 4
Not completed — Lost to Follow-up | 3
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | BeneFactor IX (BeneFIX)
Number analyzed (Participants) | 35
Age Continuous [Mean (Standard Deviation); unit: Years] | 25.7 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 35

OUTCOME MEASURES:

1. Primary Outcome: Investigator Hemostatic Efficacy Assessment of Participants After 8 Hours Post Infusion
Description: Investigator Hemostatic Efficacy Assessment was based on response of bleeding episodes to BeneFIX treatment on 4-point rating scale: Excellent(1): definite pain relief or improvement in signs of bleeding starting within 8 hrs after infusion, with no additional infusion; Good(2): definite pain relief or improvement in signs of bleeding starting within 8 hrs or following infusion; Moderate(3): probable or slight improvement starting after 8 hours following infusion; No Response(4): no improvement at all between infusions or during 24 hour interval following an infusion, or condition worsens.
Time Frame: 8 hours post infusion
Population: FAS population included all participants who were treated and had at least 1 evaluable efficacy assessment after treatment.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | BeneFactor IX (BeneFIX)
Number analyzed (Participants) | 34
Units on a scale | 1.70 (0.72)

2. Primary Outcome: Investigator Hemostatic Efficacy Assessment of Participants After 24 Hours Post Infusion
Description: as for outcome 1
Time Frame: 24 hours post infusion
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | BeneFactor IX (BeneFIX)
Number analyzed (Participants) | 34
Units on a scale | 1.58 (0.71)

3. Primary Outcome: Percentage of Participants With FIX Inhibitor Development
Description: Incidence of FIX inhibitor was defined as any result determined as positive at local laboratory, and confirmed at central laboratory with Nijmegen assay result >=0.6 Bethesda Unit (BU). Incidence was stratified by participant exposure history - Minimally Treated Patients (MTPs): those who had received at least one prior FIX infusion, and <= 100 documented Exposure Days (EDs); while Previously Treated Patients (PTPs): those who had received >100 documented prior EDs. When number of prior EDs for an individual was not known to be at least 100, participants were included in the MTP population.
Time Frame: Baseline up to 6 months
Population: Safety Set (SS) population included all enrolled participants who had taken at least 1 dose of drug.The 'n' is signifying those participants who received study drug and were evaluated for this measure at the timepoint for each visit respectively.
Measure: Number; unit: Percentage of Participants
Arm/Group | BeneFactor IX (BeneFIX)
Number analyzed (Participants) | 35
Percentage of Participants
  Total (n=35) | 2.86
  MTP (n=24) | 4.17
  PTP (n=11) | 0

4. Secondary Outcome: Number of Infusions Required to Treat Each Bleed
Description: The number of BeneFIX infusions required to treat each bleeding episode were analyzed. The average frequency of BeneFIX infusions per hemorrhage incidence to treat every hemorrhage was equal to the total number of injections throughout the study divided by total number of hemorrhagic events.
Time Frame: Baseline up to 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Infusions
Arm/Group | BeneFactor IX (BeneFIX)
Number analyzed (Participants) | 34
Infusions | 1.20 (0.86)

5. Secondary Outcome: FIX Incremental Recovery
Description: FIX recovery was assessed by evaluating FIX:C after initial exposure and following 6 months of repeated exposures to BeneFIX. A modified FIX recovery study was performed at Day 1 (Visit 2) and Month 6/Final/Early Termination visits (Visit 4) and when clinically indicated at the applicable on-demand visits. Blood samples for determination of FIX:C were collected immediately before BeneFIX infusion and at 30 minutes (±5 minutes) after the start of infusion. Post-infusion blood samples were collected via venipuncture in arm contralateral to arm used for infusion.
Time Frame: Baseline (Visit 2) up to 6 months (Visit 4)
Population: FAS population included all participants who were treated and had at least 1 evaluable efficacy assessment after treatment. The 'n' is signifying those participants who received study drug and were evaluated for this measure at the timepoint for each visit respectively.
Measure: Mean (Standard Deviation); unit: IU/dL per IU/kg
Arm/Group | BeneFactor IX (BeneFIX)
Number analyzed (Participants) | 34
IU/dL per IU/kg
  Visit 2 (n=30) | 0.760 (0.222)
  Visit 4 (n=31) | 0.727 (0.275)

6. Secondary Outcome: Percentage of Participants With Less Than Expected Therapeutic Effect (LETE)
Description: The incidence of LETE for on-demand treatment was defined as no response after each of 2 successive infusions within 24 hours for the same bleeding event in the absence of confounding factors.
Time Frame: Baseline up to 6 months
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | BeneFactor IX (BeneFIX)
Number analyzed (Participants) | 34
Percentage of Participants | 0

7. Secondary Outcome: Percentage of Participants With Allergic-Type Allergic Reactions
Description: Hypersensitivity to undesirable (damaging, discomfort-producing and sometimes fatal) reactions produced by the normal immune system. Hypersensitivity reactions require a pre-sensitized (immune) state of the host.
Time Frame: Baseline up to 6 months
Population: SS population included all enrolled participants who had taken at least 1 dose of drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | BeneFactor IX (BeneFIX)
Number analyzed (Participants) | 35
Percentage of Participants | 0

8. Secondary Outcome: Percentage of Participants With Thrombosis
Description: Thrombosis is the formation of a blood clot (thrombus) inside a blood vessel, obstructing the flow of blood through the circulatory system. When a blood vessel is injured, the body uses platelets and fibrin to form a blood clot to prevent blood loss.
Time Frame: Baseline up to 6 months
Population: SS population included all enrolled participants who had taken at least 1 dose of drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | BeneFactor IX (BeneFIX)
Number analyzed (Participants) | 35
Percentage of Participants | 0

9. Secondary Outcome: Percentage of Participants With Red Blood Cell (RBC) Agglutination
Description: RBC Agglutination is the clumping of red blood cells in the presence of an antibody. The antibody or other molecule bonded multiple particles and joined them, creating a large complex.
Time Frame: Baseline up to 6 months
Population: SS population included all enrolled participants who had taken at least 1 dose of drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | BeneFactor IX (BeneFIX)
Number analyzed (Participants) | 35
Percentage of Participants | 0

ADVERSE EVENTS:
Time Frame: From screening until 30 days after the last visit (Month 6/Final/Early Termination visit
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study.
Arm/Group | BeneFactor IX (BeneFIX)
Serious Adverse Events (participants affected / at risk) | 2/35
Other Adverse Events (participants affected / at risk) | 19/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BeneFactor IX (BeneFIX) (N=35)
Hemorrhage intracranial (Nervous system disorders) | 1 (1)
Hemophilia B with anti factor IX (Congenital, familial and genetic disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BeneFactor IX (BeneFIX) (N=35)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Inflammation (General disorders) | 2 (2)
Edema peripheral (General disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 2 (2)
Joint Sprain (Injury, poisoning and procedural complications) | 2 (2)
Alanine aminotransferase increased (Investigations) | 1 (1)
Hematocrit abnormal (Investigations) | 1 (1)
Hemoglobin abnormal (Investigations) | 1 (1)
Red blood cell count abnormal (Investigations) | 1 (1)
Vertigo (Nervous system disorders) | 1 (1)
Synovitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Hemorrhage (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.